CLINICAL TRIAL: NCT04170829
Title: A Phase Ib Study to Determine the Safety and Immunogenicity of the Candidate Middle East Respiratory Syndrome Coronavirus (MERS-CoV) Vaccine ChAdOx1 MERS in Healthy Adult Middle Eastern Volunteers
Brief Title: A Clinical Trial to Determine the Safety and Immunogenicity of Healthy Candidate MERS-CoV Vaccine (MERS002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT18/004/R; MERS002 (Other Grant/Funding Number: University of Oxford)
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Middle East Respiratory Syndrome Coronavirus
Keywords: MERS-CoV; ChAdOx1 MERS
MeSH Terms: interventions — Middle East respiratory syndrome vaccine

STUDY DESIGN:
Intervention Model Description: Open-labelled, non-randomised, dose escalation, extension for a first-in-human, single centre, phase Ib clinical trial
Masking Description: Open-labelled, non-randomised, dose escalation, extension for a first-in-human, single centre, phase Ib clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (n=6) (Experimental): will be administered ChAdOx1 MERS: 5 x 109 vp ChAdOx1 MERS
  Interventions: Biological: ChAdOx1 MERS
- Group 2 (n=9) (Experimental): will be administered ChAdOx1 MERS: 2.5 x 1010 vp ChAdOx1 MERS
  Interventions: Biological: ChAdOx1 MERS
- Group 3 (n=9) (Experimental): will be administered ChAdOx1 MERS: 5 x 1010 vp ChAdOx1 MERS
  Interventions: Biological: ChAdOx1 MERS

INTERVENTIONS:
Biological: ChAdOx1 MERS — a replication-deficient simian adenoviral vector expressing the spike (S) protein of MERS Coronavirus.

SUMMARY:
A phase Ib study to determine the safety and immunogenicity of the candidate Middle East Respiratory Syndrome Coronavirus (MERS-CoV) vaccine ChAdOx1 MERS in healthy adult Middle Eastern volunteers

DETAILED DESCRIPTION:
This is an open-label, dose escalation phase 1b trial to assess the safety and immunogenicity of the candidate ChAdOx1 MERS vaccine in healthy Middle Eastern adult volunteers aged 18-50. The first-in-human trial is now being conducted in Oxford in UK healthy adult volunteers. The vaccine will be administered intramuscularly.

Volunteers will be recruited and vaccinated at the King Abdulaziz Medical City, M-NGHA, Riyadh. There will be 3 study groups and a total of 24 volunteers will be enrolled. Staggered enrolment will apply for the first three volunteers within each group. Volunteers will be first recruited into Group 1 and subsequently into Groups 2 and 3 following interim clinical safety reviews. Volunteers will be allocated to a study group by selecting eligible volunteers for enrolment in the order in which they were deemed eligible, following screening.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy* ME adults aged 18 to 50 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to access the volunteer's medical history.
4. For females only, not planning to get pregnant during the study and a negative pregnancy test on the day(s) of screening and vaccination. Effective methods of contraception must be used. See section 6.3.3
5. Agreement to refrain from blood donation during the course of the study
6. Provide written informed consent

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data.
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
7. Any history of anaphylaxis in relation to vaccination
8. Pregnancy, lactation or willingness/intention to become pregnant during the study
9. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
10. History of serious psychiatric condition likely to affect participation in the study
11. Bleeding disorder (eg. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
12. Any other serious chronic illness requiring hospital specialist supervision
13. Suspected or known current alcohol use.
14. Suspected or known drug abuse in the 5 years preceding enrolment
15. Seropositive for hepatitis B surface antigen (HBsAg)
16. Seropositive for hepatitis C virus (antibodies to HCV)
17. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
19. History of exposure to MERS-CoV *
20. History of contact with camels. Defined as working in farms or barns; having been within 6 feet (2 meters) of a sick camel without PPE; or consumption of raw milk or uncooked meat. For this study, 30 days prior to screening will be considered.
21. History of allergic reaction to Aminoglycoside antibiotics. *rRT-PCR testing of nasopharyngeal specimen , at the discretion of PI, may be indicated when a volunteer is suspected to be asymptomatic carrier.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited local and systemic adverse events | 28 days following the vaccination
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. Change from baseline for safety laboratory measures will also be collected. Occurrence of serious adverse events will be collected during the whole study duration

SECONDARY OUTCOMES:
Measures of immunogenicity to the ChAdOx1 MERS vaccine | 6.5 months following completion of the vaccination regimen
  ELISA to quantify antibodies to MERS Spike protein antigen Ex vivo ELISpot responses to MERS Spike protein antigen

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bosaeed, MD, Principal Investigator — Ministry of National Guard-Health Affairs (MNGHA)
Locations (1):
- King Abdulaziz Medical City, National Guard Health Affairs, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosaeed M, Balkhy HH, Almaziad S, Aljami HA, Alhatmi H, Alanazi H, Alahmadi M, Jawhary A, Alenazi MW, Almasoud A, Alanazi R, Bittaye M, Aboagye J, Albaalharith N, Batawi S, Folegatti P, Ramos Lopez F, Ewer K, Almoaikel K, Aljeraisy M, Alothman A, Gilbert SC, Khalaf Alharbi N. Safety and immunogenicity of ChAdOx1 MERS vaccine candidate in healthy Middle Eastern adults (MERS002): an open-label, non-randomised, dose-escalation, phase 1b trial. Lancet Microbe. 2022 Jan;3(1):e11-e20. doi: 10.1016/S2666-5247(21)00193-2. Epub 2021 Nov 3. PMID 34751259